CLINICAL TRIAL: NCT02722005
Title: The Impact of Family Financial Support on Health Related Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Adam Schickedanz, Clinical Instructor in Pediatrics and Clinical Scholar, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UCLASchickedanzFCHRQOL
Record Dates: First submitted 2016-03-24; First posted 2016-03-29 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Quality of Life; Socioeconomic Status
Keywords: Health related quality of life; Financial Coaching; Medical Financial Partnership; Social Determinants of Health; Socioeconomic status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Financial Coaching & Access to Services (Experimental): Enrollment in one-to-one financial coaching intervention to support savings, income, and credit while reducing debt using available tools in the community development field.
  Interventions: Behavioral: Financial Coaching; Behavioral: Access to referral to social services
- Access to Services (Active Comparator): Participants will have access to a host of referrals to social services (this is the intervention for this group)
  Interventions: Behavioral: Access to referral to social services

INTERVENTIONS:
Behavioral: Financial Coaching — One-to-one financial coaching focused on credit, debt, savings, and income supports.
  Arms: Financial Coaching & Access to Services
Behavioral: Access to referral to social services — Access to referral to a host of social services.

SUMMARY:
The investigators have partnered with financial coaching organizations to establish what the investigators have termed a "Medical-Financial Partnership (MFP)" that offers financial coaching to improve financial and mental health. The investigators will evaluate the MFP's impact on health related quality of life using the Patient Reported Outcome Measurement Information System (PROMIS) 10 Global Short Form.

DETAILED DESCRIPTION:
Financial coaching is a new tool in the field of community development, but it has already demonstrated significant financial impact in a number of studies, including one randomized trial conducted by the Urban Institute. Financial coaching improves participant financial literacy, budgeting, saving for financial emergencies, and debt level. The investigators' project will help clinicians and the field of community economic development understand health and well-being through a new economic lens and assess the health-related impacts of the emerging field of financial coaching. The investigators have partnered with financial coaching organizations to establish what they have termed a "Medical-Financial Partnership (MFP)" that offers financial coaching to improve financial and mental health. The investigators will evaluate the MFP's impact on health related quality of life using the Patient Reported Outcome Measurement Information System (PROMIS)10 Global Short Form.

Community-based participants will be recruited from South Los Angeles and randomized to receive either monthly financial coaching plus access to referral for social services (intervention) or access to referral for social services alone (control). Inclusion criteria include having dependents under age 18, having some form of income, and having a tax identification number (social security number or Individual Tax Identification Number). Participants will be surveyed quarterly regarding their health related quality of life using the PROMIS-10 Global Short Form.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be caregivers/parents with one or more child dependents, some form of income, and a tax identification number.

Exclusion Criteria:

* Inability to participate in financial coaching due to activity/cognitive limitations or primary language other than English or Spanish.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-03; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Health-Related Quality of Life | Up to one year (if possible)
  We will assess differences between the groups and over time in terms of health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Adam Schickedanz, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- LIFT-LA in Affiliation with UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Participant consents do not include data sharing beyond the study and there exists no appropriate repository for data sharing.